CLINICAL TRIAL: NCT01106508
Title: A Phase I, Multi-center, Open Label, Dose Escalation Study of LEQ506, an Oral Smoothened Inhibitor, in Patients With Advanced Solid Tumors
Brief Title: A Dose Finding and Safety Study of Oral LEQ506 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEQ506X2101; 2009-017969-30 (EudraCT Number)
Record Dates: First submitted 2010-04-16; First posted 2010-04-20 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2016-01

CONDITIONS: Advanced Solid Tumors; Recurrent or Refractory Medulloblastoma; Locally Advanced or Metastatic Basal Cell Carcinoma
Keywords: Advanced solid tumors; recurrent or refractory medulloblastoma; locally advanced or metastatic basal cell carcinoma; hedgehog pathway inhibitor
MeSH Terms: conditions — Recurrence; Medulloblastoma; Carcinoma, Basal Cell | interventions — NVP-LEQ506

ARMS (1):
- LEQ506 (Experimental)
  Interventions: Drug: LEQ506

INTERVENTIONS:
Drug: LEQ506

SUMMARY:
This first-in-human dose-escalation study is to characterize the safety, tolerability, pharmacokinetics and pharmacodynamics of LEQ506 given orally on a daily dosing schedule in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of advanced solid tumor, recurrent or refractory medulloblastoma or locally advanced or metastatic basal cell carcinoma)
* Protocol defined laboratory parameters
* Performance status ≤ 2
* Patients must have fully recovered from the prior effects of major surgery and from any acute toxicities of prior chemotherapy/radiotherapy

Exclusion Criteria:

* History of central nervous system tumors of symptomatic brain metastases (excludes medulloblastoma patients)
* Impairment of gastrointestinal function or unresolved nausea, vomiting or diarrhea
* Impairment of cardiac function or significant cardiac disease
* Pregnant or lactating women
* Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose and characterize the dose limiting toxicities of LEQ506 | 21 day cycles

SECONDARY OUTCOMES:
To characterize the safety and tolerability of LEQ506 treatment | 21 day cycles
To characterize the pharmacokinetics of LEQ506 | 21 day cycles
To characterize the pharmacodynamic effects of LEQ506 in skin and tumor samples | 21 day cycles
Tumor response | every 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (2):
  - University of California at Los Angeles UCLA LeConte Location, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Novartis Investigative Site, Utrecht, Netherlands
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Oxford, United Kingdom

REFERENCES:
- See also: Results for CLEQ506X2101 on the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14808